CLINICAL TRIAL: NCT03602144
Title: Breakfast, Energy Metabolism, and Skeletal Muscle Health in Obese Children
Brief Title: Breakfast and Muscle Health in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Jamie Baum, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BEMS1
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Body Weight Changes; Body Composition; Muscle Mass; Energy Expenditure; Nutrition
MeSH Terms: conditions — Body Weight Changes | interventions — Carbohydrates; Proteins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate (Active Comparator): Participants will receive a carbohydrate-based smoothie every morning for 6 weeks (42 days).
  Interventions: Other: Carbohydrate
- Protein (Experimental): Participants will receive a protein-based smoothie every morning for 6 weeks (42 days).
  Interventions: Other: Protein

INTERVENTIONS:
Other: Carbohydrate — Participants will receive a carbohydrate-based breakfast beverage everyone morning for 42 days.
  Arms: Carbohydrate
Other: Protein — Participants will receive a protein-based breakfast beverage everyone morning for 42 days.
  Arms: Protein

SUMMARY:
One in every three children ages 2-19 years is overweight or obese. Although multifactorial in nature, obesity is primarily attributed to a mismatch between energy intake and energy expenditure (EE). Daily EE (DEE) can be partitioned between resting metabolic rate (RMR), EE associated with physical activity, and the thermic effect of food (TEF). RMR corresponds to the energy needed to sustain the body functions at rest and is also related to body composition (i.e., ratio of skeletal muscle mass to fat mass). Skeletal muscle mass is a large contributor to RMR; the more skeletal muscle mass, the higher the RMR (i.e., more energy expended at rest). In addition, muscle plays a central role in whole body protein metabolism and disrupted muscle metabolism is associated with the development of many common chronic diseases associated with obesity such as type 2 diabetes and cardiovascular disease. Although the contribution of disrupted muscle metabolism to chronic disease is well-established in older adults, the potential impact in children is unknown. The overall objective for this primary project application is to determine the role of breakfast protein consumption in improving energy metabolism, energy balance and skeletal muscle health in obese, school-aged children.

ELIGIBILITY:
Inclusion Criteria:

* Resides within Northwest Arkansas
* Age 8-12 years old
* BMI >5th percentile
* All ethnicities

Exclusion Criteria:

* Food allergies
* Dietary restrictions
* Regularly skip breakfast (> 5 times per week)
* Prescription medications
* Claustrophobic
* Fear of needles
* Classified as a picky eater by parent/guardian

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Whole body energy expenditure (WBEE) | WBEE will be measured as the change between WBEE during day 1 and day 42 of the intervention.
  WBEE will be measured using doubly labeled water.

SECONDARY OUTCOMES:
Appetite (VAS) | VAS will be measured on day 1 and day 42.
  Appetite response to test beverages will be measured using visual analog scales. Appetite and palatability were assessed using a traditional 100-mm visual analog scale (VAS) [33] with opposing anchors (e.g., "extremely hungry" or "not hungry at all") at time points 0, 15, 30, 60, 90, and 120 min. Questions consisted of: "how hungry do you feel at this moment", "how full do you feel at this moment", "how strong is your desire to eat this moment" and "how much food do you think you can eat at this moment". A higher number is associated with increased hunger.
Glycemic Response | Glycemic response will be measured on day 1 and day 42.
  Glucose and insulin will be measured using commercially available kits.
Muscle mass | Change in muscle mass will be determined by the difference in muscle mass between day 1 and day 42.
  Muscle mass will be measured using stable isotope-labeled creatine.
Muscle fractional synthesis rate (FSR) | FSR will be determined as the change between baseline (day 0) and day 42.
  FSR will be measured using deuterated water and markers of muscle health in plasma.
Whole body protein turnover (WPT) | Change in WPT will be determined by the difference in WPT between day 1 and day 42.
  WPT will be measured via stable isotope-labeled nitrogen.
Resting energy expenditure (REE) | Change in REE will be determined by the difference in REE between day 1 and day 42.
  REE will be measured using indirect calorimetry.
Body composition | Change in body composition will be determined by the difference in body composition between day 1 and day 42.
  Body composition will be measured via dual x-ray absorptiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie I Baum, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States